CLINICAL TRIAL: NCT00436618
Title: Phase II Trial of Everolimus (RAD001) in Relapsed/Refractory Lymphoma
Brief Title: Everolimus in Treating Patients With Lymphoma That Has Relapsed or Not Responded to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC048G; P30CA015083 (NIH); MC048G (Other: Mayo Clinic Cancer Cancer); 1042-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2018-10

CONDITIONS: Leukemia; Lymphoma; Lymphoproliferative Disorder
Keywords: recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; small intestine lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent grade 3 follicular lymphoma; recurrent marginal zone lymphoma; refractory chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; recurrent adult diffuse large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent mantle cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; post-transplant lymphoproliferative disorder; recurrent adult diffuse small cleaved cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoproliferative Disorders; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Relapsed aggressive non-Hodgkin lymphoma (Experimental): Study 1. Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
  Interventions: Drug: Everolimus
- Relapsed indolent non-Hodgkin lymphoma (Experimental): Study 2. Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
  Interventions: Drug: Everolimus
- Uncommon lymphomas (Experimental): Study 3. Includes Hodgkin's lymphomas. Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
  Other Names: Mayo abbreviation: RAD001

SUMMARY:
RATIONALE: Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

PURPOSE: This phase II trial is studying the side effects and how well everolimus works in treating patients with lymphoma that has relapsed or not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the tumor response in patients with relapsed or refractory indolent non-Hodgkin lymphoma (closed to accrual as of 8/18/08), aggressive non-Hodgkin's lymphoma (closed to accrual as of 2/7/08 except for diffuse large B cell lymphoma, grade III follicular lymphoma, or transformed lymphoma), or uncommon lymphoma (closed to accrual as of 9/2/08), including Hodgkin's lymphoma, treated with everolimus.

Secondary

* Evaluate overall survival, progression-free survival, and time to disease progression in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to histology (aggressive lymphoma [closed to accrual as of 2/7/08 except for diffuse large B cell lymphoma, grade III follicular lymphoma, or transformed lymphoma] vs indolent lymphoma [closed to accrual as of 8/18/08] vs uncommon lymphoma [closed to accrual as of 9/2/08]).

Patient receive oral everolimus daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and tissue collection at baseline and periodically during study treatment for translational research studies. Blood and tissue samples are analyzed for biomarkers to study the effect of everolimus on lymphoma.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven* relapsed or refractory lymphoma, including the following:

  * Aggressive lymphoma (closed to accrual as of 2/7/08 except for diffuse large B cell lymphoma, grade III follicular lymphoma, or transformed lymphoma)

    * Transformed lymphoma
    * Diffuse large B-cell lymphoma
    * Mantle cell lymphoma
    * Grade 3 follicular lymphoma
    * Precursor B-cell lymphoblastic leukemia/lymphoma
    * Mediastinal (thymic) large B-cell lymphoma
    * Burkitt's lymphoma/leukemia
    * Precursor T-cell lymphoblastic leukemia/lymphoma
    * Primary cutaneous anaplastic large cell lymphoma
    * Primary systemic type anaplastic large cell lymphoma
  * Indolent lymphoma (closed to accrual as of 8/18/08)

    * Small lymphocytic lymphoma/chronic lymphocytic leukemia
    * Grade 1 or 2 follicular lymphoma
    * Extranodal marginal zone B-cell lymphoma of MALT type
    * Nodal marginal zone B-cell lymphoma
    * Splenic marginal zone B-cell lymphoma
  * Uncommon lymphoma (closed to accrual as of 9/2/08)

    * Unspecified peripheral T-cell lymphoma
    * Anaplastic large cell lymphoma (T and null cell type)
    * Lymphoplasmacytic lymphoma (Waldenstrom's macroglobulinemia)
    * Central Nervous System (CNS) lymphoma
    * Post-transplant lymphoproliferative disorder
    * Mycosis fungoides/Sezary syndrome
    * Hodgkin's lymphoma
    * Primary effusion lymphoma
    * Blastic Natural Killer(NK)-cell lymphoma
    * Adult T-cell leukemia/lymphoma
    * Nasal type extranodal NK/T-cell lymphoma
    * Enteropathy type T-cell lymphoma
    * Hepatosplenic T-cell lymphoma
    * Subcutaneous panniculitis-like T-cell lymphoma
    * Angioimmunoblastic T-cell lymphoma

NOTE: *Biopsies performed < 6 months prior to study entry are allowed; biopsy-proven CNS lymphoma (at any time) does not require a re-biopsy in order to be eligible for this study

* Previously treated disease

  * Patients with aggressive lymphoma (closed to accrual as of 8/24/07) OR Hodgkin's lymphoma must have received or be ineligible for potentially curative therapy, including stem cell transplantation
* Measurable disease** by CT scan or MRI, defined by 1 of the following:

  * At least 1 unidimensionally measurable lesion > 2 cm in diameter

    * Skin lesions may be used if they meet this criterion and are photographed with a ruler
  * More than 5,000/mm³ tumor cells in the blood

NOTE: **For patients with lymphoplasmacytic lymphoma without measurable lymphadenopathy, measurable disease may be defined by bone marrow lymphoplasmacytosis with > 10% lymphoplasmacytic cells or aggregates, sheets, lymphocytes, plasma cells, or lymphoplasmacytic cells on bone marrow biopsy AND quantitative Immunoglobulin M(IgM) monoclonal protein > 1,000 mg/dL

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group(ECOG) performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 8 g/dL
* Total bilirubin ≤ 2 times upper limit of normal (ULN) OR direct bilirubin ≤ 1.5 times ULN
* aspartate aminotransferase(AST) ≤ 3 times ULN (5 times ULN if liver involvement is present)
* Creatinine ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to provide blood samples and portion of bone marrow aspirate and biopsy during study participation
* Able to swallow intact study medication tablets
* No other life-threatening illness (unrelated to tumor)
* No serious non-malignant disease (e.g., active infection or other condition) that, in the opinion of the investigator, would preclude study participation
* No other active malignancy requiring treatment or that would preclude study participation
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior myelosuppressive chemotherapy or biologic therapy (unless the patient has recovered from the nadir of the previous treatment)
* More than 3 weeks since prior radiotherapy (unless the acute side effects associated with therapy are resolved)
* Concurrent stable (i.e., not increased within the past month) chronic doses of corticosteroids, with a maximum dose of 20 mg of prednisone per day, is allowed if prescribed for disorders other than lymphoma (e.g., rheumatoid arthritis, polymyalgia rheumatica, adrenal insufficiency, or asthma)

  * Non-escalating doses of steroids at the lowest possible dosing level are allowed for CNS lymphoma
* No other concurrent investigational ancillary therapy
* No other concurrent chemotherapy, immunotherapy, or radiotherapy
* No concurrent participation in any other clinical trial involving a pharmacologic agent (e.g., drugs, biologics, immunotherapy, or gene therapy) for symptom control or therapeutic intent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Result] Ghobrial IM, Gertz M, Laplant B, Camoriano J, Hayman S, Lacy M, Chuma S, Harris B, Leduc R, Rourke M, Ansell SM, Deangelo D, Dispenzieri A, Bergsagel L, Reeder C, Anderson KC, Richardson PG, Treon SP, Witzig TE. Phase II trial of the oral mammalian target of rapamycin inhibitor everolimus in relapsed or refractory Waldenstrom macroglobulinemia. J Clin Oncol. 2010 Mar 10;28(8):1408-14. doi: 10.1200/JCO.2009.24.0994. Epub 2010 Feb 8. PMID 20142598
- [Result] Johnston PB, Inwards DJ, Colgan JP, Laplant BR, Kabat BF, Habermann TM, Micallef IN, Porrata LF, Ansell SM, Reeder CB, Roy V, Witzig TE. A Phase II trial of the oral mTOR inhibitor everolimus in relapsed Hodgkin lymphoma. Am J Hematol. 2010 May;85(5):320-4. doi: 10.1002/ajh.21664. PMID 20229590
- [Result] Witzig TE, Reeder CB, LaPlant BR, Gupta M, Johnston PB, Micallef IN, Porrata LF, Ansell SM, Colgan JP, Jacobsen ED, Ghobrial IM, Habermann TM. A phase II trial of the oral mTOR inhibitor everolimus in relapsed aggressive lymphoma. Leukemia. 2011 Feb;25(2):341-7. doi: 10.1038/leu.2010.226. Epub 2010 Dec 7. PMID 21135857
- [Result] Zent CS, LaPlant BR, Johnston PB, Call TG, Habermann TM, Micallef IN, Witzig TE. The treatment of recurrent/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL) with everolimus results in clinical responses and mobilization of CLL cells into the circulation. Cancer. 2010 May 1;116(9):2201-7. doi: 10.1002/cncr.25005. PMID 20166206
- [Derived] Witzig TE, Reeder C, Han JJ, LaPlant B, Stenson M, Tun HW, Macon W, Ansell SM, Habermann TM, Inwards DJ, Micallef IN, Johnston PB, Porrata LF, Colgan JP, Markovic S, Nowakowski GS, Gupta M. The mTORC1 inhibitor everolimus has antitumor activity in vitro and produces tumor responses in patients with relapsed T-cell lymphoma. Blood. 2015 Jul 16;126(3):328-35. doi: 10.1182/blood-2015-02-629543. Epub 2015 Apr 28. PMID 25921059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 277 patients were accrued from 4 medical clinics in the United States between August 2005 and May 2010. One patient withdrew before starting treatment and thus excluded from the results.
Groups:
- Relapsed Aggressive Non-Hodgkin Lymphoma: Study 1.
  Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
  Everolimus : Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
- Relapsed Indolent Non-Hodgkin Lymphoma: Study 2.
  Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
  Everolimus : Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
- Uncommon Lymphomas: Study 3. Includes Hodgkin's lymphomas.
  Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
  Everolimus : Everolimus 10 mg orally daily for 4 week cycle. Repeat until progression, unacceptable toxicity, refusal, or alternative therapy at any time.
Period: Overall Study
Arm/Group | Relapsed Aggressive Non-Hodgkin Lymphoma | Relapsed Indolent Non-Hodgkin Lymphoma | Uncommon Lymphomas
Started | 114 | 55 | 107
Completed | 84 | 28 | 46
Not Completed | 30 | 27 | 61
Not completed — Withdrawal by Subject | 5 | 8 | 11
Not completed — Adverse Event | 8 | 8 | 9
Not completed — Alternate Treatment | 3 | 4 | 12
Not completed — Other Medical Problems | 3 | 1 | 7
Not completed — Death | 4 | 2 | 3
Not completed — New Primary or Other Reasons | 6 | 2 | 12
Not completed — Still on treatment | 1 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relapsed Aggressive Non-Hodgkin Lymphoma | Relapsed Indolent Non-Hodgkin Lymphoma | Uncommon Lymphomas | Total
Number analyzed (Participants) | 114 | 55 | 107 | 276
Age, Continuous [Median (Full Range); unit: years] | 70 [36 to 92] | 67 [33 to 85] | 60 [20 to 85] | 66 [20 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 25 | 28 | 94
  Male | 73 | 30 | 79 | 182
Region of Enrollment [Number; unit: participants]
  United States | 114 | 55 | 107 | 276
Hodgkin versus Non-Hodgkin Lymphoma [Number; unit: participants]
  Hodgkin Lymphoma | 0 | 0 | 29 | 29
  Non-Hodgkin Lymphoma | 114 | 55 | 78 | 247

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response, Defined by Disease: Chronic Lymphocytic Leukemia(CLL): Clinical Complete or Complete or Nodular Partial or Partial Remission, Waldenstrom: Complete or Partial Response, All Others: Complete or Complete Unconfirmed or Partial Response.
Description: CLL (subset of patients in the Relapsed Indolent Non-Hodgkin Lymphoma group): 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100000/μL platelets, >11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions.
  Waldenstrom (subset of patients in the Uncommon Lymphomas group): >50% reduction in serum immunoglobulin M(IgM) levels (by serum protein electrophoresis (SPEP)) during any point while in this study, and no appearance of new lesions.
  All others: at least a 50% decrease in the sum of the products of the greatest diameters (SPD) of the six largest dominant nodes or nodal masses and no increase in the size of other nodes, liver, or spleen and splenic and hepatic nodules must regress by at least 50% in the SPD and no new sites of disease.
Time Frame: 5 years
Population: 276 out of 277 were analyzed for response. One patient was excluded because of patient refusal before starting treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients in group
Arm/Group | Relapsed Aggressive Non-Hodgkin Lymphoma | Relapsed Indolent Non-Hodgkin Lymphoma | Uncommon Lymphomas
Number analyzed (Participants) | 114 | 55 | 107
percentage of patients in group | 26 [19 to 35] | 35 [22 to 49] | 49 [39 to 58]

2. Secondary Outcome: Overall Survival
Description: The overall survival or survival time is defined as the time from registration to death due to any cause. The distribution of overall survival was estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Relapsed Aggressive Non-Hodgkin Lymphoma | Relapsed Indolent Non-Hodgkin Lymphoma | Uncommon Lymphomas
Number analyzed (Participants) | 114 | 55 | 107
years | 0.66 [0.44 to 0.99] | 2.45 [1.04 to 4.97] | 3.41 [2.31 to 5.13]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration to the time of progression or death due to any cause. Progression-free survival was estimated using the method of Kaplan-Meier.
  Progression is defined as the following:
  CLL (subset of patients in the Relapsed Indolent Non-Hodgkin Lymphoma group): >=50% increase in nodes from nadir or >=50% increase in liver/spleen size from nadir.
  Waldenstrom (subset of patients in the Uncommon Lymphomas group): >50% lymph node increase in SPD of > 1 node or new nodes, or >50% liver/spleen size increase, or > 25% IgM (by SPEP) increase, or lymphocyte morphology transformation to a more aggressive histology.
  All Others: New lesions or >=50% lymph nodes.
Time Frame: 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Relapsed Aggressive Non-Hodgkin Lymphoma | Relapsed Indolent Non-Hodgkin Lymphoma | Uncommon Lymphomas
Number analyzed (Participants) | 114 | 55 | 107
years | 0.18 [0.16 to 0.27] | 0.60 [0.41 to 1.03] | 0.79 [0.52 to 1.09]

4. Secondary Outcome: Time to Progression
Description: The time to progression is defined as the time from registration to the time of progression. The distribution of time to progression was estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Relapsed Aggressive Non-Hodgkin Lymphoma | Relapsed Indolent Non-Hodgkin Lymphoma | Uncommon Lymphomas
Number analyzed (Participants) | 114 | 55 | 107
years | 0.18 [0.16 to 0.29] | 0.60 [0.42 to 1.16] | 0.90 [0.62 to 1.49]

ADVERSE EVENTS:
Arm/Group | Relapsed Aggressive Non-Hodgkin Lymphoma | Relapsed Indolent Non-Hodgkin Lymphoma | Uncommon Lymphomas
Serious Adverse Events (participants affected / at risk) | 38/114 | 11/55 | 25/107
Other Adverse Events (participants affected / at risk) | 113/114 | 55/55 | 107/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed Aggressive Non-Hodgkin Lymphoma (N=114) | Relapsed Indolent Non-Hodgkin Lymphoma (N=55) | Uncommon Lymphomas (N=107)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 5 (6)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (5) | 4 (4)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (5) | 3 (3) | 2 (2)
Platelet count decreased (Investigations) | 15 (17) | 5 (7) | 12 (18)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed Aggressive Non-Hodgkin Lymphoma (N=114) | Relapsed Indolent Non-Hodgkin Lymphoma (N=55) | Uncommon Lymphomas (N=107)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 107 (426) | 49 (207) | 103 (770)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (4) | 1 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 37 (57) | 22 (48) | 41 (93)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (16) | 8 (11) | 21 (27)
Nausea (Gastrointestinal disorders) | 33 (46) | 17 (22) | 35 (54)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 26 (31) | 7 (8) | 21 (29)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 4 (7) | 1 (8) | 4 (18)
Fatigue (General disorders) | 34 (42) | 21 (22) | 32 (63)
Fever (General disorders) | 8 (8) | 2 (2) | 1 (1)
General symptom (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Visceral edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cecal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 6 (6) | 9 (11)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (3)
Sinusitis (Infections and infestations) | 2 (3) | 2 (2) | 4 (5)
Skin infection (Infections and infestations) | 7 (8) | 2 (2) | 4 (5)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1) | 7 (10)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (2) | 2 (4)
Viral hepatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (5)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 5 (12)
Aspartate aminotransferase increased (Investigations) | 8 (12) | 3 (3) | 2 (7)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (3) | 0 (0) | 5 (5)
Leukocyte count decreased (Investigations) | 70 (190) | 25 (78) | 67 (285)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 62 (106) | 25 (58) | 51 (148)
Platelet count decreased (Investigations) | 91 (380) | 40 (177) | 74 (375)
Serum cholesterol increased (Investigations) | 12 (21) | 6 (13) | 7 (16)
Weight loss (Investigations) | 4 (4) | 1 (2) | 5 (14)
Anorexia (Metabolism and nutrition disorders) | 9 (10) | 3 (3) | 4 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 27 (45) | 8 (19) | 15 (31)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 14 (24) | 7 (13) | 9 (25)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (4) | 5 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4) | 6 (6)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Accessory nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (6) | 1 (1) | 4 (6)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (25) | 0 (0) | 4 (4)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (4) | 9 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (4) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 8 (11) | 5 (6) | 13 (15)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (6)
Hypertension (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes